CLINICAL TRIAL: NCT03859830
Title: Clinical Observation of the Performance of Artis Dialysis System, ArtiSet PrePost and Ultra HDF Line in Treatments of Patients With End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXU012184
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artis Dialysis System (Experimental): One midweek HDF session for a duration of 4 hours.
  Interventions: Device: Artis Dialysis System, ArtiSet PrePost and Ultra HDF Line
- AK200 Ultra S (Active Comparator): One midweek HDF session for a duration of 4 hours.
  Interventions: Device: AK200 Ultra S, extracorporeal circulation conduct of blood purification

INTERVENTIONS:
Device: Artis Dialysis System, ArtiSet PrePost and Ultra HDF Line — The HDF session will be performed in post-dilution volume-controlled mode, with a minimum target total convective volume (VCtot) of 16 L and blood flow rate (QB) set at 200-300 mL/min.
  Arms: Artis Dialysis System
Device: AK200 Ultra S, extracorporeal circulation conduct of blood purification — The HDF session will be performed in post-dilution volume-controlled mode, with a minimum target total convective volume (VCtot) of 16 L and blood flow rate (QB) set at 200-300 mL/min.
  Arms: AK200 Ultra S

SUMMARY:
The incidence and prevalence of chronic kidney disease are increasing worldwide, as is the number of patients progressing to End-Stage Renal Disease (ESRD). China has experienced an increased accessibility and affordability of dialysis treatment, which in turn has brought about an increase in the number of patients receiving Renal Replacement Therapy (RRT).Without RRT, either in the form of maintenance dialysis or transplantation, ESRD is fatal.

The scope of the trial is to observe the performance of Artis Dialysis System, ArtiSet PrePost and Ultra HDF Line versus AK 200 Ultra S, extracorporeal circulation conduct of blood purification apparatus and Ultra Steriset as the comparator devices in treatment of patients using hemodialysis (HD) or hemodiafiltration (HDF) for ESRD.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 to ≤75 years of age with diagnosis of ESRD
* Patients on thrice weekly HD for a minimum of 3 months who received at least one 4 hour HDF treatment in the past two weeks prior to study enrollment with a total convection volume (VCtot) (including UF) of equal or greater than 16 L post-dilution
* Body weight (BW) ≥ 40 Kg
* Patients with stable dialysis profiles:

  1. Kt/Vurea ≥ 1.2 which is taken within 4 weeks before study enrollment
  2. Dialysis prescription stable over 6 recent treatments
* Patients on stable anticoagulation dose
* Patients who have an adequate arteriovenous fistula (AVF) or graft, capable of providing a QB with 200-300 mL/min range
* Patients able to give informed consent (IC) after an explanation of the proposed study
* Patients who receive in-center treatment HD at a site that routinely implements high flux dialysis and/or HDF

Exclusion Criteria:

* Patients who are human immunodeficiency virus (HIV) positive, or with active Hepatitis A (HAV), Hepatitis B (HBV) or Hepatitis C (HBC)
* Patients with known hemodynamic instability, bleeding risks and coagulation disorders
* Patients with active or ongoing infection
* Patients with advanced liver, heart or pulmonary disease, as judged by the Investigator, that would not be suitable for participation in the study
* Patients with any comorbidity possibly conflicting with the study purpose or procedures as judged by the Investigator
* Patients who are currently participating in other interventional clinical trials or have participated in another interventional clinical trial within one (1) month of the current study that may interfere with this study as judged by the Investigator.
* Pregnant women, lactating women and women or men who plan to have a baby and refuse to apply the effective contraceptive methods during the study period
* Patients with active cancer
* Patients who have acute renal failure
* Patients who are pre-scheduled for a living kidney transplant within the next two months, who plan a change to PD within the next two months, or who require single needle dialysis therapy
* Patients diagnosed with New York Heart Association (NYHA) Class IV congestive heart failure, or acute coronary syndrome and/or who have suffered a myocardial infarction within the three months prior to the start of the study
* Patients with a history of severe mental disorders
* Patients who have had an allergic response to polyarylethersulfone or polysulfone membrane

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
Number of participants successfully completing HDF without interruption of therapy during Dialysis | Day 1 (One Midweek HDF Treament Session, 4 hour duration)
  Defined as participants not having an interruption in therapy for greater than 15 continuous minutes due to a technical reason of all the enrolled patients in the same group. If there is more than one interruption due to technical reasons, the criteria for failure should be the sum of all interruptions being greater than 15 minutes.
Number of Participants by Level of Effectiveness of Disposable Tubing during and after Dialysis | Day 1 (One Midweek HDF Treament Session, 4 hour duration)
  Participant recorded as "yes" or "no" by categories of (1) blood flow in the tubing is smooth without obstruction, blood flow rate meets requirement of the patient's hemodialysis prescription and finish the dialysis procedure, the (2) connections are free from blood and air leakage and detachment, (3) there is no folding, cracking or rupture in tubing during dialysis procedure.
Reduction ratio of β2-Microglobulin during and after Dialysis | Day 1 (One Midweek HDF Treament Session, 4 hour duration)

SECONDARY OUTCOMES:
Single-pool Kt/V urea during and after Dialysis | Day 1 (One Midweek HDF Treament Session, 4 hour duration)
  Computing formula: spKt/V = -ln (R - 0.008t) + (4 - 3.5R) x (ΔBW/BW). Where R is the blood urea after hemodialysis/ blood urea before hemodialysis; t is time in hours; ΔBW is the weight change values after hemodialysis, namely ultrafiltration volume in liters; BW is weight in kilograms.
Urea Reduction Ratio (URR) during and after Dialysis | Day 1 (One Midweek HDF Treament Session, 4 hour duration)
Number of Participants by Level of Appearance of Disposable Tubing during and after Dialysis | Day 1 (One Midweek HDF Treament Session, 4 hour duration)
  Participants with tubing as flexible, transparent, and smooth (it is easy to observe the presence of bubbles) recorded categorically as "yes" or "no."
Number of Participants by Level of Elasticity of Pump Lines during and after Dialysis | Day 1 (One Midweek HDF Treament Session, 4 hour duration)
  Participants with the blood and fluid lines showing good elasticity and good resilience after being rolled without obvious deformity after dialysis recorded categorically as "yes" or "no."

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Investigational Site, Beijing, Beijing Municipality
  - Investigational Site, Foshan, Guangdong
  - Investigational Site, Wuhan, Hubei
  - Investigational Site, Nanjing, Jiangsu
  - Investigational Site, Shenyang, Liaoning
  - Investigational Site, Hangzhou, Zhejiang
  - Investigational Site, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No